CLINICAL TRIAL: NCT06207253
Title: The Antimicrobial Potential of Diclofenac Sodium as an Intracanal Medicament During Root Canal Treatment: A Randomized Clinical Trial
Brief Title: The Antimicrobial Potential of Diclofenac Sodium as an Intracanal Medicament
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: British University In Egypt (Other)
Responsible Party: Principal Investigator, Summer Elsayed, Principle Investigator, British University In Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23-039
Record Dates: First submitted 2023-12-14; First posted 2024-01-16 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Endodontic Disease; Pulp Disease, Dental; Intracanal Medication
Keywords: Sodium diclofenac; Intracanal medication; Calcium hydroxide; Apical periodontitis
MeSH Terms: conditions — Dental Pulp Diseases; Periapical Periodontitis | interventions — Diclofenac; Calcium Hydroxide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- High concentration of diclofenac sodium (Experimental): High concentration of diclofenac sodium mixed with saline
  Interventions: Drug: Diclofenac Sodium
- Low concentration of diclofenac sodium (Active Comparator): Low concentration of diclofenac sodium mixed with saline
  Interventions: Drug: Diclofenac Sodium
- Calcium hydroxide (Active Comparator): Calcium hydroxide paste form
  Interventions: Drug: Calcium hydroxide

INTERVENTIONS:
Drug: Diclofenac Sodium — placement of intracanal medication for the three groups will be done after cleaning and shaping of the root canals and it will be left for one week.
  Arms: High concentration of diclofenac sodium; Low concentration of diclofenac sodium
Drug: Calcium hydroxide — placement of intracanal medication for the three groups will be done after cleaning and shaping of the root canals and it will be left for one week.
  Arms: Calcium hydroxide

SUMMARY:
The goal of this randomized clinical trial is to evaluate the capability of the material to exert bacterial reduction of diclofenac sodium versus of that calcium hydroxide paste when these materials are used as intracanal medications in permanent molar teeth with chronic apical periodontitis.

The main question[s] it aims to answer are:

• Will the diclofenac sodium (NSAIDs) possess antimicrobial efficacy to be used effectively as an intracanal medicament similar to that of calcium hydroxide in primary endodontic treatment? Participants will be allocated randomly into three equal groups by using computer generated randomization, according to the type of intracanal medication.

DETAILED DESCRIPTION:
The aim of the present study is to evaluate the capability of the material to exert bacterial reduction of diclofenac sodium versus of that calcium hydroxide paste when these materials are used as intracanal medications in permanent molar teeth with chronic apical periodontitis. The evaluation is to be done using quantitative microbiological assessment from samples extracted from root canals before and after intracanal medicament placement in roots of permanent molars, having PAI score ≥ 2.

ELIGIBILITY:
Inclusion Criteria:

* Patients with teeth diagnosed with apical periodontitis
* Periapical Index (PAI) ≥ 2
* The teeth are restorable

Exclusion Criteria:

* Teeth with immature roots
* Non restorable teeth
* Medically compromised patients with systemic complication that would alter the treatment.
* Teeth with internal/external root resorption
* Patient with an allergy to diclofenac sodium

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Bacterial count | On the seventh day from of intracanal medication placement appointment
  Variation in bacterial count in high concentration of Diclofenac Sodium group compared by group of low concentration of Diclofenac Sodium group and calcium hydroxide group.

SECONDARY OUTCOMES:
Periapical healing | participants will be recalled after 6 months from the obturation for radiographic examination.
  Change in the size of periapical lesion (according to Periapical index scale). The participants will be recalled after at least 6 months, and radiographic examination of the treated tooth will be performed. Preoperative and recall radiographs of teeth will be each assigned a Periapical index score by 2 blinded, independent, and calibrated examiners according to periapical index score (PAI):
  PAI 1: Normal periapical structure. PAI 2: Bone structural changes indicating but not pathognomonic for apical periodontitis.
  PAI 3: Bone structural changes with some mineral loss characteristic for apical periodontitis.
  PAI 4: Well-defined apical radiolucency. PAI 5: Radiolucency with radiating expansion of bone structural changes.
incidence and intensity of pain | Pain intensity will be assessed at 24 hours, 48 hours and 72 hours following initial treatment using a visual analogue scale
  Patient will receive visual analogue scale (VAS) that will include a 10 cm line in which number 0 will correspond to no pain and number 10 will indicate unacceptable pain. Evaluation of intensity and incidence of pain, will be assessed each day for the following first three days after intracanal placement appointment (after 24 hours, 48 hours and 72 hours).
Incidence of flare-ups | Presence of flare-ups will be recorded each day after the intracanal medication placement visit till the next visit (after seven days).
  Flare-up will be defined to patients as the development of swelling after treatment and will be represented by "Yes" (flare-up) or "No" (no flare-up). It will be recorded on chart that will given to the patients after the initial treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Shehab Eldin M Saber, doctoral, Study Director — british university in Egypt- dentistry collage
Locations (1):
- British university in Egypt, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No